CLINICAL TRIAL: NCT05466318
Title: ChiCGB Versus BEAM With Autologous Stem-Cell Transplantation in High-risk Hodgkin and Non-Hodgkin Lymphoma - A Prospective, Multi-centered, Randomized Clinical Trial
Brief Title: ChiCGB vs BEAM in High-risk or R/R Lymphomas
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Principle Investigator, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCGB 2.0
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cladribine; Gemcitabine; Busulfan; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChiCGB (Experimental): Treated with chidamide, cladribine, gemcitabine and busulfan(ChiCGB) therapy followed by autologous hematopoietic stem cell transplantation.
  Interventions: Drug: Chidamide; Drug: Cladribine; Drug: Gemcitabine; Drug: Busulfan; Procedure: Autologous hematopoietic stem cell transplant
- BEAM (Active Comparator): Treated with BCNU, etoposide, cytarabine and melphalan (BEAM) therapy followed by autologous hematopoietic stem cell transplantation.
  Interventions: Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Procedure: Autologous hematopoietic stem cell transplant

INTERVENTIONS:
Drug: Chidamide — 30 mg oral twice weekly for 2 weeks
  Arms: ChiCGB
Drug: Cladribine — 6 mg/m2 intravenously once daily @ Day -7 ~ -3
  Arms: ChiCGB
Drug: Gemcitabine — 2500 mg/m2 intravenously @ Day -7, -3
  Arms: ChiCGB
Drug: Busulfan — 3.2 mg/kg intravenously once daily @ Day -7 ~ -4
  Arms: ChiCGB
Drug: Carmustine — 300 mg/m2 intravenously @ Day -8
  Arms: BEAM
Drug: Etoposide — 200 mg/m2 intravenously once daily @ Day -7 ~ -4
  Arms: BEAM
Drug: Cytarabine — 400 mg/m2 intravenously once daily @ Day -7 ~ -4
  Arms: BEAM
Drug: Melphalan — 140 mg/m2 intravenously @ Day -3
  Arms: BEAM
Procedure: Autologous hematopoietic stem cell transplant — autologous hematopoietic stem cells infusion after ChiCGB or BEAM chemotherapy

SUMMARY:
High-dose chemotherapy (HDT) with autologous stem cell transplantation (ASCT) plays a vital role in treating high-risked or relapsed/refractory lymphoma. Our previous study showed chidamide combined with cladribine, gemcitabine, and busulfan (ChiCGB) as conditioning therapy improved the survival of these patients. So we designed this trial to verify if ChiCGB were better than BCNU, etoposide, cytarabine, and melphalan (BEAM). Patients with diffuse large B cell or extra-nodal NK/T cell Lymphoma who consent to this study will be randomized into the trial group who receive ChiCGB or the control group whom receive BEAM. Patients will be followed for up to 2 years after the hematopoietic cell transplantation (HCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary refractory or recurrent diffuse large B cell lymphoma or extra-nodal NK/T cell lymphoma that do not qualify for treatment protocols of higher priority.
* Relapsed patients should respond to 2nd or 3rd line salvage chemotherapy and attain at least partial response before recruitment.
* Adequate renal function, as defined by estimated serum creatinine clearance >/=50 ml/min and/or serum creatinine </= 1.8 mg/dL.
* Adequate hepatic function, as defined by serum glutamate oxaloacetate transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) </= 3 x upper limit of normal; serum bilirubin and alkaline phosphatase </= 2 x upper limit of normal.
* Adequate pulmonary function with forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusing capacity of lung for carbon monoxide (DLCO) >/= 50% of expected corrected for hemoglobin.
* Adequate cardiac function with left ventricular ejection fraction >/= 50%. No uncontrolled arrhythmias or symptomatic cardiac disease.
* Performance status 0-1. 10. Negative Beta diffusing capacity of the lung for carbon monoxide (HCG) text in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization

Exclusion Criteria:

* Central nervous system lymphoma
* Patients relapsed after autologous stem cell transplantation
* Bone marrow was involved by lymphoma
* Patients with active hepatitis B or C(HBV DNA >/=10,000 copies/mL).
* Active infection requiring parenteral antibiotics
* HIV infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and a normal cluster of differentiation 4 (CD4) counts
* Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.
* Patients with a corrected QT interval(QTc) longer than 500 ms

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Progression free survival of this group of patients at the end of 2 year

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival of this group of patients at the end of 2 year
100 day adverse events (AE) | 100 days from transplant
  non-hematologic adverse events @ Day +100
100 day complete response (CR) rate | 100 days from transplant
  Complete response @ Day +100

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - People's Hospital of Deyang City, Deyang, Deyang
  - Chengdu Third People's Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Chengdu First People's Hospital, Chengdu, Sichuan
  - PLA Western Theater Command General Hospital, Chengdu, Sichuan
  - Dazhou Central Hospital, Dazhou, Sichuan
  - Southwest Medical University, Luzhou, Sichuan
  - Central Hospital of Mianyang City, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Zigong First People's Hospital, Zigong, Sichuan
  - Guangyuan Central Hospital, Guangyuan, Sihcuan

IPD SHARING:
Plan to Share IPD: Yes
Release after the publication of results of this trial
Supporting Information: Study Protocol
Time Frame: after the publication of results of this trial